CLINICAL TRIAL: NCT04915118
Title: NT-proBNP Assessment in a HFrEF Population in Germany
Brief Title: A Study Called NATION-OS to Learn About the Link Between N-terminal proBNP (NT-proBNP) Levels and Medical Problems Due to Heart Failure (HF) in German Patients With HF
Acronym: NATION-OS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21868
Record Dates: First submitted 2021-05-11; First posted 2021-06-07 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure (HF)
MeSH Terms: conditions — Heart Failure | interventions — Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with HFrEF: Patients with HFrEF (Heart failure with reduced ejection fraction) who had a previous decompensation event.
  Interventions: Other: Decompensation event

INTERVENTIONS:
Other: Decompensation event — NT-proBNP (N-terminal pro B-type natriuretic) peptide distribution in patients with HFrEF who had a previous decompensation event.
  Other Names: Biomarker

SUMMARY:
Researchers are looking for a better way to treat heart failure (HF), a condition in which the heart does not pump blood as well as it should.

Research has shown that the levels of a hormone called N-terminal proBNP (NT-proBNP) in the body can be used for differential diagnosing of HF. NT-proBNP is released by the heart when there is an increase in heart pressure. The levels of NT-proBNP can indicate whether medical problems are likely to happen due to HF. These medical problems are called "decompensation events." The higher a person's NT-proBNP levels is expected, the higher their risk of developing HF and having decompensation events.

So, the researchers in this study want to learn about NT-proBNP levels and decompensation events in German patients with a common type of HF called heart failure with reduced ejection fraction (HFrEF). In patients with HFrEF, the muscle on the left chamber of the heart does not pump blood as well as it should. The researchers will collect information from patients and their health records for about 300 adult patients in Germany with HFrEF who have been receiving standard of care treatment for their condition. Standard of care treatments are treatments that doctors commonly use to treat patients.

The researchers will study and record the levels of NT-proBNP levels and any changes in the health of the patients at time of NT-proBNP measurement.

The researchers will collect this information between May 2021 and September 2021.

The patients in this study :

* have had any HF-decompensation event since January 2016
* have had at least 1 NT-proBNP measurement done before the study

The researchers will collect the following information about the patients:

* the results of NT-proBNP measurements
* the date of the NT-proBNP measurements
* the number and type of decompensation events

ELIGIBILITY:
Inclusion Criteria:

* Female or male patient, aged 18 years or older at the time of HF diagnosis
* Diagnosis of heart failure with reduced ejection fraction confirmed by echocardiography
* Patient on HFrEF standard of care treatment with guideline-based therapy
* One or more HF decompensation(s) within observation period defined as HFH or the need for IV diuretic treatment
* Signed informed consent if patient is alive at start of data collection
* At least one NT-proBNP value available prior enrollment, fulfilling the below criteria:

  * NT-proBNP value was assessed in an outpatient setting exactly at 01-JAN-2016 or later
  * NT-proBNP value was assessed and within six months after a decompensation event within observational period.
  * At time of NT-proBNP measurement patients need to be hemodynamically stable without signs of residual congestion

Exclusion Criteria:

At time of NT-proBNP measurement

* Participation in an investigational program with interventions outside of routine clinical practice
* Awaiting heart transplantation or has/anticipates receiving an implanted ventricular assist device
* Has acute coronary syndrome (unstable angina, non-ST elevation myocardial infarction, or ST elevation myocardial infarction) or coronary revascularization (coronary artery bypass grafting or percutaneous coronary intervention) Estimated glomerular filtration rate (eGFR) calculated based on the Modification of Diet in Renal Disease (MDRD) equation < 15 ml/min/1.73m2 or chronic dialysis
* Severe hepatic insufficiency (CHILD Pugh C)
* Acute inflammatory disease
* Malignancy
* Treatment with Vericiguat (which may be available to patients in Germany in Q3 2021 but not at time of protocol development)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be collected for patients who had at least one available NT-proBNP value in the past, that was assessed in an outpatient setting exactly at 01 JAN-2016 or later and within six months after a decompensation event.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Proportion of NT-proBNP < 5314pg/ml | within 6 months after decompensation event
  Range of NT-proBNP values and the proportion of NT-proBNP < 5314pg/ml in patients with HFrEF who had a previous decompensation event.
  The first NT-proBNP value, will be described via summary statistics, as well as by a frequency table based on categorized NT-proBNP values. The summary statistics as well as the proportion of patients within different NT-proBNP categories (i.e. </>=5314pg/ml) will be presented overall and stratified by number of decompensation event during observation period.
Range of NT-proBNP values | within 6 months after decompensation event
  Range of NT-proBNP values and the proportion of NT-proBNP < 5314pg/ml in patients with HFrEF who had a previous decompensation event.
  The first NT-proBNP value, will be described via summary statistics, as well as by a frequency table based on categorized NT-proBNP values. The summary statistics as well as the proportion of patients within different NT-proBNP categories (i.e. </>=5314pg/ml) will be presented overall and stratified by number of decompensation event during observation period.

SECONDARY OUTCOMES:
Range of NT-proBNP values across demographic characteristics | within 6 months after decompensation event
  Demographic characteristics will be described by frequency tables and/or summary statistics. The patients´ medical history conditions will be displayed by a frequency table. Patients with specific prior and concomitant medication will be presented by frequency tables.
  The standard of care for heart failure treatment (including Beta Blocker, Diuretics, ACEi or ARB, MRA, Sacubitril/Valsartan, ICD, Biventricular Pacemaker) will be tabulated by patient frequencies.
Range of NT-proBNP values across clinical patient characteristics | within 6 months after decompensation event
  Patient characteristics (e.g. comorbidities, HFH, NYHA class) will be described by frequency tables and/or summary statistics. The patients´ medical history conditions will be displayed by a frequency table. Patients with specific prior and concomitant medication will be presented by frequency tables.
  The standard of care for heart failure treatment (including Beta Blocker, Diuretics, ACEi or ARB, MRA, Sacubitril/Valsartan, ICD, Biventricular Pacemaker) will be tabulated by patient frequencies.

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.